CLINICAL TRIAL: NCT06911476
Title: From Inflammation Biomarkers to Remoddeling (FAPI PET/CT) Towards Personalized Diagnosis in Post-acute Sequelae of COVID-19
Brief Title: From Inflammation to Remodelling Towards Personalized Diagnosis in Post-acute Sequelae of COVID-19
Acronym: LIBERATE
Status: Not yet recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor
Other Study IDs: 19097; ZonMW (Other Grant/Funding Number: 10430172310012); 2024-511294-29-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-01; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: PASC Post Acute Sequelae of COVID 19; Long COVID; Long Covid-19; PASC; FAPI; FAP; Fibroblast Activation Protein Inhibitor; Fibroblast; Restrictive Lung Disease
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, nose brushes and muscle biopsies that will be analysed via single cell RNA (scRNA) analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Former PASC patients: Former PASC patients or healthy controls. Fatigue Severity Scale ≥ 4 at time of inclusion
- PASC patients: PASC patients with persistent dyspnea and fatigue. Fatigue Severity Scale ≤ 4 at time of [68Ga]FAPI PET/CT after having previously recorded score of ≥ 4 or equivalent.
- Back-up cohort - 'healthy' controls: Patients without self-reported complaints and past SARS-CoV-2 infection (which would have resulted in a Fatigue Severity Scale ≤ 4) or without experienced confirmed SARS-CoV-2 infection.

SUMMARY:
Rationale: The diagnosis and pathogenesis of long COVID remains unknown. We have previously shown that [68Ga]FAPI Positron Emission Tomography-Computed Tomography (PET/CT) imaging shows potential for diagnosis and molecular understanding of this syndrome. We have previously shown that fibroblast activation protein (FAP) can be imaged in the lung, muscle and nasopharynx of long COVID patients (with dyspnea and fatigue). However, these preliminary data are derived from a selective group of patients with long COVID after critical COVID-19. We aim to explore the generalizability of these findings in patients with long COVID with dyspnea and fatigue, irrespective of the severity of their acute SARS-CoV-2 infection.

Primary objective: To assess if pulmonary fibroblast activity, measured by [68Ga]FAPI-46 PET/CT, is higher in patients with current long COVID dyspnea and fatigue compared to patients with resolved complaints.

Study design: This is a ZonMw funded single centre prospective observational cohort study of long COVID-19 patients with dyspnea and fatigue.

Study population: We will recruit 60 adult long COVID patients (aged >20 years) of which 30 have complaints of dyspnea and fatigue and compare them to 30 patients with resolved complaints and healthy controls.

Main study parameters/endpoints: The primary endpoint is FAP expression in the lung measured by [68Ga]FAPI-46 PET/CT. Secondary endpoints are the expression of FAP in other tissues (muscle) and the relation between FAP and inflammation and remodelling biomarkers in various biological samples (e.g. serum/nasal epithelium).

Study procedures: In a single visit day the following data and samples will be collected: questionnaires, a lung function test, 6-minute walking test, blood samples, nose swabs, [68Ga]FAPI PET/CT scan and HRCT scan. When increased [68Ga]FAPI uptake is measured in the muscles a muscle biopsy will be performed as well.

ELIGIBILITY:
Inclusion Criteria:

- Self-reported complaints of dyspnea or fatigue > 3 months after SARS-CoV-2 infection confirmed with PCR, serology test or COVID-19 Reporting and Data System (CO-RADS) score 4/5.

Exclusion Criteria:

* Inability or unwilling to give informed consent.
* History of claustrophobia or feeling of inability to tolerate supine position for the PET/CT scans.
* Individuals who are pregnant or currently breastfeeding are not eligible to participate

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the P4O2 COVID-19 cohort (The Netherlands - www.p4o2.org). If too few patients from the P4O2 cohort are willing or eligible to participate in the LIBERATE study, 'healthy' controls from other cohorts may be included as a third control group to meet the required number of participants.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pulmonary FAP expression | Day 1
  To compare pulmonary FAP expression between patients with persistent PASC and patients recovered from PASC. Pulmonary FAP expression will be measured via the pulmonary FAPI uptake on the [68Ga]FAPI-46 PET/CT scan. Uptake is measured as whole lung SULmean (standardized uptake value corrected for lean body mass) corrected for the background signal (bloodpool). Resulting in the target-to-background ratio (TBR) of the whole lung.

SECONDARY OUTCOMES:
Whole body FAP expression | Day 1
  To compare whole body FAPI uptake in patients with persistent PASC vs patients recovered from PASC. Whole body FAPI uptake is measured in the muscle via automated segmentation. Mean muscle uptake values are calculated.
Pulmonary FAP expression vs clinical endpoints | Day 1
  To compare pulmonary FAPI uptake (expressed as the mean of the whole lung) to clinical endpoints (e.g. lung function, 6-minute walking test (6-MWT) and self-reported daily impairments assessed by several questionnaires).
Whole body FAP expression vs clinical endpoints | Day 1
  To compare whole body FAPI uptake (expressed as the mean of the whole lung) to clinical endpoints (e.g. 6-minute walking test (6-MWT) and self-reported daily impairments assessed by several questionnaires).
Serum biomarkers | Day 1
  To explorer serum biomarkers (e.g. soluble FAP and cytokines/growthfactors) and cellular phenotypes of inlammation and remodelling in relation to FAPI uptake (expressed as TBRmean of the whole lung).

OTHER OUTCOMES:
HRCT vs pulmonary FAP expression | Day 1
  Visual assessment of HRCT abnormalities matching pulmonary FAPI uptake.
Muscle biopsies | Day 1
  Patients willing to give additional informed consent for a muscle biopsy will be evaluated for increased muscle FAPI uptake (SUVmax of >4.5). In these patients an ultrasound guided muscle biopsy will be performed of a high uptake area (>4.5 SUV) and a low uptake area (<4 SUV). Tissue examination as well as single cell RNA analysis will be performed to explorer the relation between FAP expression and activated remoddeling programs.

CONTACTS AND LOCATIONS:
Overall Officials: J Pillay, MD PhD, Principal Investigator — Department of Intensive Care, University Medical Center Groningen

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available upon reasonable request